CLINICAL TRIAL: NCT06033404
Title: Registry of Patients Undergoing Anesthesia or Intensive Care Maneuvers
Brief Title: Anesthesia and Critical Care Registry
Acronym: ARIA
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Other Study IDs: ARIA - 40/INT//2023
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Normal Clinical practice — Normal Clinical practice

SUMMARY:
In recent decades, knowledge in the anesthesiology field has increasingly expanded, allowing for the refinement of monitoring techniques, therapies, and local-regional anesthesia maneuvers, and for the extension of care to a larger number of patients, including those previously excluded due to advanced age or comorbidities. Similarly, Intensive care management has continuously evolved, following innovations in the field of drugs and with the great diffusion of extracorporeal supports. The fundamental importance of registry studies has been recognized in this context to rapidly generate reliable data and improve the quality of care.

This prospective observational study is aimed at collecting data of all patients (expected 300,000) undergoing anesthesia or intensive care maneuvers at our institution. This registry aims to assist in carrying out registry-based clinical studies focused on improving current therapeutic and patient management standards.

DETAILED DESCRIPTION:
The study aims to collect data on 300,000 patients who undergo anesthesia and/or resuscitation procedures at the IRCCS San Raffaele Scientific Institute over a 10 years period. The information collected will include demographic data, anthropometric data, past and/or current clinical history of the patient, anamnestic clinical-instrumental data related to the anesthetic activity, data on therapeutic measures taken during stay in intensive care units, laboratory parameters, diagnostic tests, therapeutic procedures carried out during hospitalization, patient satisfaction, and evaluation scales. All this data will be anonymized prior insertion in the database, with the aim of creating a registry that can be used for scientific research. This registry aims to assist in carrying out registry-based clinical studies focused on improving current therapeutic and patient management standards. The duration of observation of each patient will be variable, depending on the length of hospital stay and/or the duration of the diagnostic-therapeutic process. The analysis will follow the clinical course of patients from admission to hospital discharge, with the possibility of conducting telephone follow-ups for certain categories of patients after 1 year. Statistical analyses will be performed by grouping or describing patients based on their characteristics or in relation to the type of anesthetic and resuscitation procedures they undergo.

This study will follow the ethical principles outlined in the Helsinki Declaration and the current regulations for Observational Studies. All patients will be fully informed about the aspects of the study and their written informed consent will be required before participation.

Participation in the study is voluntary and free. No additional costs are expected for data collection and analysis: given the observational nature of the study, insurance coverage is not required.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Anesthesia or Critical care
* Signed informed consent.

Exclusion Criteria:

Refused informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients undergoing Anesthesia or critical care -related maneuvers admitted to our hospital. All patients will follow their normal course of diagnosis/treatment without any further requirements for the scope of this study other than those provided in the normal management of patients with this condition. Furthermore, any decision regarding drug or procedure will be made by the physician based on her/his clinical judgment in the context of clinical practice, independently from the decision to include the patient in this study. No follow-up medical and/or imaging examinations/laboratory analysis after hospital discharge are needed by the present study design.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes of patients urdergoing anesthesia and/or critical care | hospital discharge (usually <=30 days)
  This study will collect data on the anesthesia-related and hospital outcome of patients undergoing anesthesia and intensive care. Due to the large sample size and heterogeneity of populations, further analysis will be planned to address homogenenous subgroups of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele di Milano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lanier WL. A three-decade perspective on anesthesia safety. Am Surg. 2006 Nov;72(11):985-9; discussion 1021-30, 1133-48. doi: 10.1177/000313480607201101. PMID 17120937
- [Background] Desmarais P, Herrmann N, Alam F, Choi S, Avramescu S. Future Directions for Geriatric Anesthesiology. Anesthesiol Clin. 2019 Sep;37(3):581-592. doi: 10.1016/j.anclin.2019.05.002. Epub 2019 Jun 14. PMID 31337487
- [Background] Belletti A, Palumbo D, Zangrillo A, Fominskiy EV, Franchini S, Dell'Acqua A, Marinosci A, Monti G, Vitali G, Colombo S, Guazzarotti G, Lembo R, Maimeri N, Faustini C, Pennella R, Mushtaq J, Landoni G, Scandroglio AM, Dagna L, De Cobelli F; COVID-BioB Study Group. Predictors of Pneumothorax/Pneumomediastinum in Mechanically Ventilated COVID-19 Patients. J Cardiothorac Vasc Anesth. 2021 Dec;35(12):3642-3651. doi: 10.1053/j.jvca.2021.02.008. Epub 2021 Feb 6. PMID 33678544
- [Background] Liau A, Havidich JE, Onega T, Dutton RP. The National Anesthesia Clinical Outcomes Registry. Anesth Analg. 2015 Dec;121(6):1604-10. doi: 10.1213/ANE.0000000000000895. PMID 26579661
- [Background] Shapiro FE, Jani SR, Liu X, Dutton RP, Urman RD. Initial results from the National Anesthesia Clinical Outcomes Registry and overview of office-based anesthesia. Anesthesiol Clin. 2014 Jun;32(2):431-44. doi: 10.1016/j.anclin.2014.02.018. PMID 24882129
- [Background] Beane A, Salluh JIF, Haniffa R. What intensive care registries can teach us about outcomes. Curr Opin Crit Care. 2021 Oct 1;27(5):537-543. doi: 10.1097/MCC.0000000000000865. PMID 34393177
- [Background] Arabi YM, Azoulay E, Al-Dorzi HM, Phua J, Salluh J, Binnie A, Hodgson C, Angus DC, Cecconi M, Du B, Fowler R, Gomersall CD, Horby P, Juffermans NP, Kesecioglu J, Kleinpell RM, Machado FR, Martin GS, Meyfroidt G, Rhodes A, Rowan K, Timsit JF, Vincent JL, Citerio G. How the COVID-19 pandemic will change the future of critical care. Intensive Care Med. 2021 Mar;47(3):282-291. doi: 10.1007/s00134-021-06352-y. Epub 2021 Feb 22. PMID 33616696
- [Background] James A, De Jong A, Jeanmougin T, Blanie A, Figueiredo S, Goffin P, Le Guen M, Kantor E, Cipriani F, Campion S, Raux M, Jaber S, Futier E, Constantin JM; Societe Francaise d'Anesthesie Reanimation (SFAR) Research Network. Characteristics and outcomes of patients undergoing anesthesia while SARS-CoV-2 infected or suspected: a multicenter register of consecutive patients. BMC Anesthesiol. 2022 Feb 14;22(1):46. doi: 10.1186/s12871-022-01581-0. PMID 35164679
- [Background] Monaco F, Belletti A, Bove T, Landoni G, Zangrillo A. Extracorporeal Membrane Oxygenation: Beyond Cardiac Surgery and Intensive Care Unit: Unconventional Uses and Future Perspectives. J Cardiothorac Vasc Anesth. 2018 Aug;32(4):1955-1970. doi: 10.1053/j.jvca.2018.03.031. Epub 2018 Mar 20. PMID 29709436
- [Background] Kelly FE, Fong K, Hirsch N, Nolan JP. Intensive care medicine is 60 years old: the history and future of the intensive care unit. Clin Med (Lond). 2014 Aug;14(4):376-9. doi: 10.7861/clinmedicine.14-4-376. PMID 25099838